CLINICAL TRIAL: NCT04432129
Title: Integrated Mental Health Care and Vocational Rehabilitation Intervention to Individuals on Sick Leave Due to Anxiety, Depression, Personality Disorders, Stress and Functional Disorders
Brief Title: Integrated Mental Health Care and Vocational Rehabilitation to People With to Common Mental Disorders
Acronym: IBBIS II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amager Hospital (Other)
Collaborators: The Danish Agency for Labour Market and Recruitment (Other); Central Denmark Region (Other); Aarhus Kommune (Other); Københavns Kommune (Other)
Responsible Party: Principal Investigator, Lene Falgaard Eplov, Head of Research, Associate professor, Amager Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Version 3.1. 27.5.2020
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Common Mental Disorders; Depression; Anxiety; Personality Disorders; Functional Disease Present; Stress
Keywords: Vocational rehabilitation; Mental health services; Return to Work
MeSH Terms: conditions — Depression; Anxiety Disorders; Personality Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBBIS II (Experimental): Integrated Mental Health Care and Vocational Rehabilitation
  Interventions: Behavioral: IBBIS II
- Service As Usual (Active Comparator): Standard vocational rehabilitation and treatment
  Interventions: Behavioral: Service as Usual

INTERVENTIONS:
Behavioral: IBBIS II — The IBBIS-II service consists of:
  1. Mental health assessment.
  2. Planned integrated service. The participant has the same employment specialists and care manager throughout the intervention. A joint plan is made with shared decisions between the participant, the employment specialist and the care manager. There is a focus on disclosure (openness about illness) and involvement of relatives and significant others.
  3. Vocational rehabilitation. Focus on return to work with ongoing assessment of job goals, competencies and need of support. Participants receive help in contacting existing employers (employed) and potential employers (unemployed). Unemployed participants are offered an individualized job search effort. The focus is on competitive jobs within the community.
  4. Treatment consists of stepped care with structured treatment guidelines.
  5. When the participant has obtained work the team continues to offer support.
  Arms: IBBIS II
Behavioral: Service as Usual — Service as usual consists of standard mental health care and vocational rehabilitation
  Arms: Service As Usual

SUMMARY:
The purpose of this study is to investigate the efficacy of an integrated mental health care and vocational rehabilitation intervention for people on sick leave because of depression, stress, anxiety, personality- and functional disorders in Denmark

DETAILED DESCRIPTION:
Background:

Mental illness has an estimated financial burden on the Danish economy of 3.4 % of Gross National Product every year due to lost productivity, social benefits and healthcare costs and approximately 50 % of people receiving long-term sickness benefits have a common mental illness. Furthermore, a significant treatment gap exists where less than 30% were treated for their mental illness.

Objective:

The primary objective of the randomized trial is to examine whether people on sick leave with a diagnosis of anxiety, depression, stress, personality disorders or functional disorders, return to work faster and have a higher job retention if they receive an integrated and optimized vocational rehabilitation and mental health care intervention, compared to people who receive the standard mental health care and vocational rehabilitation service.

Method:

The trial is designed as an randomized, two-group parallel, assessor-blinded, multisite trial. A total of 800 participants with a common mental illness will randomly be assigned into two groups 1) IBBIS II, consisting of an integrated mental health care and vocational rehabilitation; or 2) Service as usual, at two sites in Denmark. The primary outcome is difference between the two groups in time to return to work at 12 months.

Results/discussion:

This study will contribute with new knowledge on vocational recovery and integrated vocational and health care interventions in a Scandinavian context.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria

* Anxiety, depression, stress, personality disorder or functional disorder diagnosed at a structured diagnostic interview based on the Mini International Neuropsychiatric Interview conducted by the IBBIS team
* Sickness benefit recipient at baseline; on sick leave from job or unemployed for a minimum of four weeks
* Resident in Copenhagen or Aarhus municipalities
* Speak sufficient Danish to participate in interviews and complete questionnaires without an interpreter
* Aged 18 or older
* Has given informed written consent

Exclusion Criteria:

* Pregnant
* High degree of suicidal ideation
* Dementia
* Abuse of alcohol or other drugs to the degree that participation in therapy is not possible
* A need for mental health treatment in secondary sector care
* Unstable somatic condition that is too severe for participation in the project
* The participant will not refrain from participating in other psychotherapeutic treatment outside the IBBIS project if the participant will be allocated to the experimental group

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Return to work | 12 months
  Difference between the two groups in time to return to work from baseline until 12 months after baseline measured whit register based data. Time to return to work is defined as a minimum of four weeks of continuous work without receiving sickness benefit.

SECONDARY OUTCOMES:
Work at one point during follow-up | 12 months
  Proportion in unsupported competitive work at 6 and 12-months follow up
Return to work | 6 months
  Time to return to work from baseline until 6 months after baseline measured whit register based data
Supported work at one point during follow-up | 12 months
  Proportion in supported work at 6 and 12-months follow up
Weeks of work | 12 months
  Number of weeks in competitive employment from baseline to 6 and 12 months
Time to new sick leave | 12 months
  The duration from return to work to potential new sick leave of more than 4 weeks within the 12-month follow-up period
Income | 12 months
  Salary income from competitive employment at 6 and 12 months after baseline
Use of psychiatric services | 12 months
  Number of admissions, inpatient days and outpatient contacts at the psychiatric hospitals at 6- and 12-months follow-up
Use of somatic services | 12 months
  Number of admissions, inpatient days and outpatient contacts at the somatic hospitals at 6- and 12-months follow-up
Use of private health care | 12 months
  Number of contacts with private health care professionals under the Health Insurance

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Eplov, PhD, Principal Investigator — Mental Health Center Copenhagen
Locations (1):
- Copenhagen Research Center for Mental Health - CORE, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be publicly available due to legal restrictions from the Danish data protection agency and the European data protection regulation

REFERENCES:
- [Background] Christensen TN, Poulsen CH, Ebersbach BK, Eplov LF. Integrated mental health care and vocational rehabilitation intervention to improve return to work rates for people on sick leave due to common mental and functional disorders (IBBIS-II)-a study protocol for a randomized clinical trial. Trials. 2022 Sep 30;23(1):820. doi: 10.1186/s13063-022-06718-7. PMID 36175977
- [Derived] Christensen TN, Hjorthoj C, Poulsen CH, Ebersbach B, Eplov LF. Integrated mental health care and vocational rehabilitation intervention to improve return to work rates for people on sick leave due to common mental and functional disorders (IBBIS-II) - results from a randomized clinical trial. Nord J Psychiatry. 2025 Jan;79(1):86-95. doi: 10.1080/08039488.2024.2446362. Epub 2025 Jan 6. PMID 39760219
- See also: study protocol article — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-022-06718-7